CLINICAL TRIAL: NCT05365841
Title: Role of Epithelial Barrier Integrity in Biologic Treatment Response of Severe Asthmatics With/Out Chronic Rhinosinusitis With Nasal Polyps (CRSwNP). Can Shedding of Epithelial Barrier Proteins be Used as Biomarker in Severe Asthma With/Out CRSwNP Management?
Brief Title: Role of Epithelial Barrier Integrity in Biologic Treatment Response of Severe Asthmatics With/Out Chronic Rhinosinusitis With Nasal Polyps (CRSwNP).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Nikolaos Tzanakis, Professor, University of Crete
Other Study IDs: 10961[213755]
Record Dates: First submitted 2022-01-18; First posted 2022-05-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Severe Eosinophilic Asthma w/wo CRSwNP
MeSH Terms: interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Severe asthma without CRSwNP: control group; n~20 of anti-IL5 naïve severe asthmatics
  Interventions: Drug: Mepolizumab 100 MG
- Severe asthma with CRSwNP: n~40 of anti-IL5 naïve severe asthmatics
  Interventions: Drug: Mepolizumab 100 MG
- subjects CRSwNP with mild or no asthma: ~25;2nd control group

INTERVENTIONS:
Drug: Mepolizumab 100 MG — Patients with SEA eligible to receive anti-IL5 treatment, which is a biologic treatment for SEA
  Groups: Severe asthma with CRSwNP; Severe asthma without CRSwNP

SUMMARY:
Advances in understanding the pathophysiology of asthma development and severity have pointed towards a prominent role of the bronchial epithelium, especially in more chronic and severe disease. Studies suggest that airway eosinophilic inflammation in asthma is linked to epithelial injury and structural changes of the airways, co called airway wall remodeling. Together the chronic airway inflammation and remodeling are associated with bronchial hyperresponsiveness, fixed airflow obstruction or progressive loss of lung function and clinical severity of asthma. Chronic rhinosinusitis with nasal polyps (CRSwNP), is another respiratory inflammatory disease often co-existing with severe asthma, sharing similar pathophysiology. The investigators hypothesize that epithelial barrier integrity may play a role in the pathophysiology of severe eosinophilic asthma and nasal polyposis and in response to anti-IL5 therapy of severe asthmatics, and that shedding of epithelial barrier proteins may be used as biomarker in the management of severe asthma. In order to study that, the investigators will conduct a prospective cohort study of adult severe asthmatics with/out CRSwNP, who live on the island of Crete, Greece and who meet the criteria for entering anti-IL5 treatment, as assessed by pulmonologist. The participants will be recruited with a convenience sampling in a period of 2 years, under real life conditions, and will be followed up for 1 year after treatment initiation. A control group of subjects diagnosed with nasal polyposis without severe asthma will be used. Eligible subjects will undergo clinical assessment with radiological (CT) and endoscopic investigations. Samples of serum, sputum, nasal secretions, as well as nasal and bronchial biopsies will be obtain for assessing clinicopathological differences among the 3 groups but also response to anti-IL5 therapy in SEA w/o CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed written consent (study participation informed consent form): Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Anti-IL5/IL5R naïve
* Confirmed asthma diagnosis and severity and treatment requirements (for severe asthma group see boxes 1-3). For the 2nd control group, patients with CRSwNP must have a diagnosis of mild asthma (GINA steps 1-2) or no asthma by pulmonologist.
* Polyposis must be bilateral, to be considered as CRSwNP
* Triggers and relevant co-morbidity have been assessed and are well controlled Triggers such as active or passive smoking, beta-blockers, aspirin/NSAIDs, allergen exposure;Comorbidities such as rhinitis, obesity, GERD, OSA, VCD, depression/anxiety.
* Age: Adults ≥18 years of age
* Any smoking status
* Any ethnicity
* Be affiliated to or a beneficiary of a social security category and/health insurance.
* Gender: Male and Eligible Female. To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control for the duration of the follow up (and for 4 months after the last injection administration). A serum pregnancy test is required of all females. This test will be performed at the initial screening visit. In addition, a urine pregnancy test can be offered (optional) for all females during each scheduled treatment visit prior to the infusion of biologic product until the 1-year follow-up visit.

Laboratory abnormality: No evidence of clinically significant abnormality (other than those seen in SEA) in the haematological, biochemical or urinalysis screen at Visit 1, as judged by the investigator.

* Asthma Exacerbation: Subjects with an ongoing asthma exacerbation should have their screening and treatment initiation visit delayed until the investigator considers the subject has returned to their baseline asthma status. If the 4-week screening period (visits 1 and 1a) has elapsed, then the subject should be considered a screening failure. An exacerbation is defined as worsening of asthma requiring the use of systemic CS and/or emergency department visit, or hospitalisation. For subjects on maintenance oral corticosteroids, an exacerbation requiring oral CS is defined as the use of oral/systemic corticosteroids at least double the existing dose for at least 3 days.
* Maintenance Asthma Therapy: No changes in the dose or regimen of baseline ICS and/or additional controller medication during the screening period (except for treatment of an exacerbation).
* Maintenance CRSwNP: No changes in the dose or regimen of baseline intranasal CS and/or additional controller medication during the screening period (except for treatment of an exacerbation).
* Subjects with a previous surgery for the removal of nasal polyps are allowed to participate and will be considered as subjects with CRSwNP (with severe asthma or not). However, any subject who had at least one surgery for removal of nasal polyps, even if at study screening he/she is free of nasal polyps, cannot be considered as a subject without CRSwNP.
* Severe asthma patients must meet requirements for biologic therapy with anti-IL5 treatment (Mepolizumab)

Exclusion Criteria:

* Pregnancy
* Current exacerbation at visit 1 (repeat screening when stable). If exacerbation is lasting up until Visit 1a then exclude subject.
* Cognitive impairment preventing completion of data collection forms
* People highly dependent on medical care
* People with significant life limiting co-morbidity
* Other eosinophilic conditions (eosinophilic granulomatosis polyangiitis (Churg-Strauss syndrome), eosinophilic oesophagitis etc)
* Unilateral polyposis
* Primary diagnosis of lung disease other than asthma (chronic obstructive lung disease (COPD), asthma-COPD overlap (ACO), interstitial lung disease, sarcoidosis, bronchiectasis, cystic fibrosis, primary ciliary dyskinesia, active tuberculosis, allergic bronchopulmonary aspergillosis (ABPA))
* Current lung cancer or other blood, lymphatic or solid organ malignancy
* Autoimmune diseases of the skin, muscle-skeletal or gastrointestinal system needing systemic corticosteroids, immunosuppressants or biologic treatment as well as individuals with granulomatosis with polyangiitis (Wegener's granulomatosis)
* Inability to attend study and treatment visits
* Inability to understand and speak Greek or English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with severe eosinophilic asthma, naive to anti-IL5/anti-IL5R treatment with or without CRSwNP who meet requirements for biologic therapy with anti-IL5 (Mepolizumab)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Differences in sputum columnar epithelial cells (CEPs) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in sputum CEPs in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  We will employ flow cytometry on freshly isolated sputum cell suspensions from participants to measure CEPs proportion and count. Previously proposed cut-off value for normal range sputum CEP proportion (CEP % high = ≥11%) or number (CEP count high = ≥18.1 × 10^4/mL) may be considered.
Differences in E-cadherin protein level in sputum and nasal secretions among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in E-cadherin protein level in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Soluble E-cadherin in sputum and nasal secretions measured with ELISA. Data will be expressed as nanograms per milliliter in original sputum/secretion. Cell surface expression of E-cadherin on columnar epithelial cells may be analyzed by flow cytometry.
Differences in nasal and bronchial epithelial thickness among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in epithelial thickness in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Epithelial thickness will be determined in biopsies by dividing the epithelial surface area by the basement membrane (BM) length
Differences in nasal and bronchial epithelial integrity among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in epithelial integrity in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Epithelial integrity will be assessed in biopsy sections and expressed as percentage (%) of BM covered with normal epithelium (a layer of basal and ciliated columnar epithelial cells without detachment from the BM)
Differences in nasal and bronchial epithelial E-cadherin expression among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in protein expression in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Epithelial E-cadherin expression in biopsies will be measure with immonohistochemistry and expressed as the percentage of BM covered with E-cadherin-positive intact epithelium and/or as strong, moderate and weak epithelial E-cadherin staining
Differences in nasal and bronchial basement membrane thickness (BM) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in Basement membrane thickness in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  BM thickness in biopsies will be expressed as BM surface area divided by BM length
Differences in CT-assessed airway wall thickness (WT) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in WT in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  We will use high resolution computer tomography of the chest to measureairway wall thickness (WT). Airway dimensions will be measured at on contiguous slices of the right apical segmental bronchus and right posterior basal segmental bronchus, from which tangential views of the bronchi can be obtained. The averaged values of the 2 bronchi will be used for analysis
Differences in CRSwNP stage among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in CRSwNP stage in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  The Lund-Mackay score is widely used in radiological staging of chronic rhinosinusitis. Although there are many scoring systems in place for sinonasal computed tomography (CT) analysis, the Lund-Mackay system has the best inter- and intraob-server agreement. In LMK scoring, the sinuses (maxillary, anterior/posterior ethmoid, sphenoid, and frontal) are each scored on a scale of 0-2 opacification (0, normal; 1, partial opacification; 2, total opacification). The ostiomeatal complex is scored on a two-point scale of 0 and 2 (0, not occluded; 2, occluded). The scores on each side ranged from 0 (complete translucency of all sinuses) to 12 (complete opacity of all sinuses), leading to a total LMK score of 24 for both sides.Of note, an aplastic (absent) frontal sinus receives a score of 0.
Differences in exacerbation rate among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in exacerbation rate in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Number of exacerbation in the past 12 months. An exacerbation is defined as worsening of asthma requiring the use of systemic CS and/or emergency department visit, or hospitalisation. For subjects on maintenance oral corticosteroids, an exacerbation requiring oral CS is defined as the use of oral/systemic corticosteroids at least double the existing dose for at least 3 days
Differences in lung function among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in lung function in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  FEV1 (liters and %predicted), FVC (liters and %predicted, FEV1/FVC (%) including pre and post bronchodilator test
Differences in need for sinus surgery among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in need for sinus surgery in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Number (%) of participants with a reduced need for sinus surgery at 1 year. Surgery will be deemed required with an ENP score of >=3, or an ENP score of 2 and a TNSS score of >7.
  Polyp (ENP) score: 0=No polyps,1=Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate, 2=Polyps reaching below the lower border of the middle turbinate, 3=Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate, 4=Large polyps causing complete obstruction of the inferior nasal cavity. The higher of the two nostril scores will be derived and used for the analysis.
  With a VAS (0 to 10 cm) the severity of 4 nasal polyposis symptoms (one VAS for each symptom): rhinorrhea; mucus in the throat; nasal blockage; loss of smell, and for total nasal symptom score (TNSS). The left-hand side of the scale (0) represents "not troublesome," and the right-hand side of the scale (10) represents "worst possible troublesome.

SECONDARY OUTCOMES:
Differences in total IgE among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in total IgE in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Total serum IgE (UI/ml)
Differences in blood eosinophil count among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in blood eosninophil count in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Blood eosinophil differential counts (number and percentage)
Differences in sputum eosinophil count among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in sputum eosinophil count in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Eosinophils count (number x10^4/mL and %) in a differential cell count obtained from induced sputum
Differences in FeNO among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in FeNO in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  Fractional Exhaled Nitric Oxide (FeNO in parts per billion)
Differences in Asthma Control Test (ACT) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in asthma control in1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  ACT includes 5 items, with 4-week recall (on symptoms and daily functioning). More specifically, ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. There is 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Differences in quality of life among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in quality of life in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  With the Asthma Quality of Life Questionnaire (AQLQ) we will assess quality of life and psychological morbidity. The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item questionnaire used to assess the physical, occupational, emotional, and social qualities of adults aged 17 to 70 years with asthma (Juniper et al, 2005).
  The AQLQ has 4 domains: symptoms (12 items), activity limitation (6 generic and 5 patient-specific items), emotional function (5 items), and environmental stimuli (4 items). The AQLQ was developed for patients exhibiting mild to moderate asthma (Aburuz et al, 2007). The AQLQ items are each scored on a 7-point Likert scale, with 1 representing maximal impairment and 7 representing no impairment. The original AQLQ includes 5 patient-specific questions in the activity limitation domain. As part of the initial interview, the patient indicates 5 activity limitations due to asthma. These 5 activity limitations are used for the remaining follow-up visits.

OTHER OUTCOMES:
Differences in Asthma Control Questionnaire (ACQ) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in asthma control in1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  ACQ has a multidimensional construct assessing symptoms (5 items--self-administred) and rescue inbronchodilator use (1 item-self-administered) with 1 week recall (for items on symptoms and rescue inhaler use), and FEV1% (1 item) completed by clinic staff. There is 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%) and scores range between 0 (totally controlled) and 6 (severely uncontrolled). ACQ >1.5 will be considered inadequately controlled asthma
Differences in CT-assessed airway wall thickness percentage (WT%) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in WT% in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  We will use high resolution computer tomography of the chest to measure the WT% calculated using the formula [WT/outer dimaeter] × 100), on contiguous slices of the right apical segmental bronchus and right posterior basal segmental bronchus, from which tangential views of the bronchi can be obtained. The averaged values of the 2 bronchi will be used for analysis
Differences in CT-assessed percentage of wall area (WA%) among 3 groups (SEA w/o CRSwNP and CRSwNP with mild or no asthma) at baseline, and change in WA% in 1-year post anti-IL5 treatment initiation in SEA w/o CRSwNP | Baseline and 1 year
  We will use high resolution computer tomography of the chest to measure the percentage of wall area (WA%) calculated using the formula [airway wall area/outer area of the bronchus] × 100), on contiguous slices of the right apical segmental bronchus and right posterior basal segmental bronchus, from which tangential views of the bronchi can be obtained. The averaged values of the 2 bronchi will be used for analysis

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - "PAGNI" University Hospital, Crete, Heraklion, Crete
  - Aikaterini Antoniou, Heraklion, Crete

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight DA, Stick SM, Hackett TL. Defective function at the epithelial junction: a novel therapeutic frontier in asthma? J Allergy Clin Immunol. 2011 Sep;128(3):557-8. doi: 10.1016/j.jaci.2011.07.031. No abstract available. PMID 21878242
- [Background] NAYLOR B. The shedding of the mucosa of the bronchial tree in asthma. Thorax. 1962 Mar;17(1):69-72. doi: 10.1136/thx.17.1.69. No abstract available. PMID 14478653
- [Background] Hoshino M, Ohtawa J. Effects of adding omalizumab, an anti-immunoglobulin E antibody, on airway wall thickening in asthma. Respiration. 2012;83(6):520-8. doi: 10.1159/000334701. Epub 2012 Jan 11. PMID 22236804
- [Background] Watelet JB, Gevaert P, Holtappels G, Van Cauwenberge P, Bachert C. Collection of nasal secretions for immunological analysis. Eur Arch Otorhinolaryngol. 2004 May;261(5):242-6. doi: 10.1007/s00405-003-0691-y. Epub 2003 Oct 9. PMID 14551791
- [Background] Lund VJ, Kennedy DW. Quantification for staging sinusitis. The Staging and Therapy Group. Ann Otol Rhinol Laryngol Suppl. 1995 Oct;167:17-21. PMID 7574265
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Background] Bousquet J, Heinzerling L, Bachert C, Papadopoulos NG, Bousquet PJ, Burney PG, Canonica GW, Carlsen KH, Cox L, Haahtela T, Lodrup Carlsen KC, Price D, Samolinski B, Simons FE, Wickman M, Annesi-Maesano I, Baena-Cagnani CE, Bergmann KC, Bindslev-Jensen C, Casale TB, Chiriac A, Cruz AA, Dubakiene R, Durham SR, Fokkens WJ, Gerth-van-Wijk R, Kalayci O, Kowalski ML, Mari A, Mullol J, Nazamova-Baranova L, O'Hehir RE, Ohta K, Panzner P, Passalacqua G, Ring J, Rogala B, Romano A, Ryan D, Schmid-Grendelmeier P, Todo-Bom A, Valenta R, Woehrl S, Yusuf OM, Zuberbier T, Demoly P; Global Allergy and Asthma European Network; Allergic Rhinitis and its Impact on Asthma. Practical guide to skin prick tests in allergy to aeroallergens. Allergy. 2012 Jan;67(1):18-24. doi: 10.1111/j.1398-9995.2011.02728.x. Epub 2011 Nov 4. PMID 22050279
- [Background] Heinzerling LM, Burbach GJ, Edenharter G, Bachert C, Bindslev-Jensen C, Bonini S, Bousquet J, Bousquet-Rouanet L, Bousquet PJ, Bresciani M, Bruno A, Burney P, Canonica GW, Darsow U, Demoly P, Durham S, Fokkens WJ, Giavi S, Gjomarkaj M, Gramiccioni C, Haahtela T, Kowalski ML, Magyar P, Murakozi G, Orosz M, Papadopoulos NG, Rohnelt C, Stingl G, Todo-Bom A, Von Mutius E, Wiesner A, Wohrl S, Zuberbier T. GA(2)LEN skin test study I: GA(2)LEN harmonization of skin prick testing: novel sensitization patterns for inhalant allergens in Europe. Allergy. 2009 Oct;64(10):1498-1506. doi: 10.1111/j.1398-9995.2009.02093.x. PMID 19772515
- [Background] Horvath I, Barnes PJ, Loukides S, Sterk PJ, Hogman M, Olin AC, Amann A, Antus B, Baraldi E, Bikov A, Boots AW, Bos LD, Brinkman P, Bucca C, Carpagnano GE, Corradi M, Cristescu S, de Jongste JC, Dinh-Xuan AT, Dompeling E, Fens N, Fowler S, Hohlfeld JM, Holz O, Jobsis Q, Van De Kant K, Knobel HH, Kostikas K, Lehtimaki L, Lundberg J, Montuschi P, Van Muylem A, Pennazza G, Reinhold P, Ricciardolo FLM, Rosias P, Santonico M, van der Schee MP, van Schooten FJ, Spanevello A, Tonia T, Vink TJ. A European Respiratory Society technical standard: exhaled biomarkers in lung disease. Eur Respir J. 2017 Apr 26;49(4):1600965. doi: 10.1183/13993003.00965-2016. Print 2017 Apr. PMID 28446552
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Coates AL, Wanger J, Cockcroft DW, Culver BH; Bronchoprovocation Testing Task Force: Kai-Hakon Carlsen; Diamant Z, Gauvreau G, Hall GL, Hallstrand TS, Horvath I, de Jongh FHC, Joos G, Kaminsky DA, Laube BL, Leuppi JD, Sterk PJ. ERS technical standard on bronchial challenge testing: general considerations and performance of methacholine challenge tests. Eur Respir J. 2017 May 1;49(5):1601526. doi: 10.1183/13993003.01526-2016. Print 2017 May. PMID 28461290
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Bulathsinhala L, Eleangovan N, Heaney LG, Menzies-Gow A, Gibson PG, Peters M, Hew M, van Boven JFM, Lehtimaki L, van Ganse E, Belhassen M, Harvey ES, Perez de Llano L, Maitland-van der Zee AH, Papadopoulos NG, FitzGerald JM, Porsbjerg C, Canonica GW, Backer V, Rhee CK, Verhamme KMC, Buhl R, Cosio BG, Carter V, Price C, Le T, Stagno d'Alcontres M, Gopalan G, Tran TN, Price D. Development of the International Severe Asthma Registry (ISAR): A Modified Delphi Study. J Allergy Clin Immunol Pract. 2019 Feb;7(2):578-588.e2. doi: 10.1016/j.jaip.2018.08.016. Epub 2018 Sep 1. PMID 30179741
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Fokkens WJ, Lund V, Bachert C, Mullol J, Bjermer L, Bousquet J, Canonica GW, Deneyer L, Desrosiers M, Diamant Z, Han J, Heffler E, Hopkins C, Jankowski R, Joos G, Knill A, Lee J, Lee SE, Marien G, Pugin B, Senior B, Seys SF, Hellings PW. EUFOREA consensus on biologics for CRSwNP with or without asthma. Allergy. 2019 Dec;74(12):2312-2319. doi: 10.1111/all.13875. Epub 2019 Jul 15. PMID 31090937
- [Background] Stevens WW, Schleimer RP, Kern RC. Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):565-72. doi: 10.1016/j.jaip.2016.04.012. PMID 27393770
- [Background] Moore WC, Bleecker ER, Curran-Everett D, Erzurum SC, Ameredes BT, Bacharier L, Calhoun WJ, Castro M, Chung KF, Clark MP, Dweik RA, Fitzpatrick AM, Gaston B, Hew M, Hussain I, Jarjour NN, Israel E, Levy BD, Murphy JR, Peters SP, Teague WG, Meyers DA, Busse WW, Wenzel SE; National Heart, Lung, Blood Institute's Severe Asthma Research Program. Characterization of the severe asthma phenotype by the National Heart, Lung, and Blood Institute's Severe Asthma Research Program. J Allergy Clin Immunol. 2007 Feb;119(2):405-13. doi: 10.1016/j.jaci.2006.11.639. PMID 17291857
- [Background] Porsbjerg C, Menzies-Gow A. Co-morbidities in severe asthma: Clinical impact and management. Respirology. 2017 May;22(4):651-661. doi: 10.1111/resp.13026. Epub 2017 Mar 22. PMID 28328160
- [Background] Radhakrishna N, Tay TR, Hore-Lacy F, Hoy R, Dabscheck E, Hew M. Profile of difficult to treat asthma patients referred for systematic assessment. Respir Med. 2016 Aug;117:166-73. doi: 10.1016/j.rmed.2016.06.012. Epub 2016 Jun 14. PMID 27492528
- [Background] Moore WC, Meyers DA, Wenzel SE, Teague WG, Li H, Li X, D'Agostino R Jr, Castro M, Curran-Everett D, Fitzpatrick AM, Gaston B, Jarjour NN, Sorkness R, Calhoun WJ, Chung KF, Comhair SA, Dweik RA, Israel E, Peters SP, Busse WW, Erzurum SC, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Identification of asthma phenotypes using cluster analysis in the Severe Asthma Research Program. Am J Respir Crit Care Med. 2010 Feb 15;181(4):315-23. doi: 10.1164/rccm.200906-0896OC. Epub 2009 Nov 5. PMID 19892860
- [Background] Shen HH, Du XF, Ying SM. [Comparison of Chinese guideline for asthma managment and prevention (2016 update) and global initiative for asthma (2017 update)]. Zhonghua Jie He He Hu Xi Za Zhi. 2018 Mar 12;41(3):166-168. doi: 10.3760/cma.j.issn.1001-0939.2018.03.003. No abstract available. Chinese. PMID 29518845
- [Background] Condreay L, Chiano M, Ortega H, Buchan N, Harris E, Bleecker ER, Thompson PJ, Humbert M, Gibson P, Yancey S, Ghosh S. No genetic association detected with mepolizumab efficacy in severe asthma. Respir Med. 2017 Nov;132:178-180. doi: 10.1016/j.rmed.2017.10.019. Epub 2017 Oct 26. PMID 29229094
- [Background] Flood-Page P, Menzies-Gow A, Phipps S, Ying S, Wangoo A, Ludwig MS, Barnes N, Robinson D, Kay AB. Anti-IL-5 treatment reduces deposition of ECM proteins in the bronchial subepithelial basement membrane of mild atopic asthmatics. J Clin Invest. 2003 Oct;112(7):1029-36. doi: 10.1172/JCI17974. PMID 14523040
- [Background] Przybyszowski M, Paciorek K, Zastrzezynska W, Gawlewicz-Mroczka A, Trojan-Krolikowska A, Orlowska A, Soja J, Pawlik W, Sladek K. Influence of omalizumab therapy on airway remodeling assessed with high-resolution computed tomography (HRCT) in severe allergic asthma patients. Adv Respir Med. 2018 Dec 30;86(6). doi: 10.5603/ARM.a2018.0046. PMID 30594995
- [Background] Samitas K, Delimpoura V, Zervas E, Gaga M. Anti-IgE treatment, airway inflammation and remodelling in severe allergic asthma: current knowledge and future perspectives. Eur Respir Rev. 2015 Dec;24(138):594-601. doi: 10.1183/16000617.00001715. PMID 26621973
- [Background] Gevaert P, Lang-Loidolt D, Lackner A, Stammberger H, Staudinger H, Van Zele T, Holtappels G, Tavernier J, van Cauwenberge P, Bachert C. Nasal IL-5 levels determine the response to anti-IL-5 treatment in patients with nasal polyps. J Allergy Clin Immunol. 2006 Nov;118(5):1133-41. doi: 10.1016/j.jaci.2006.05.031. Epub 2006 Sep 26. PMID 17088140
- [Background] Gevaert P, Calus L, Van Zele T, Blomme K, De Ruyck N, Bauters W, Hellings P, Brusselle G, De Bacquer D, van Cauwenberge P, Bachert C. Omalizumab is effective in allergic and nonallergic patients with nasal polyps and asthma. J Allergy Clin Immunol. 2013 Jan;131(1):110-6.e1. doi: 10.1016/j.jaci.2012.07.047. Epub 2012 Sep 27. PMID 23021878
- [Background] Farne HA, Wilson A, Powell C, Bax L, Milan SJ. Anti-IL5 therapies for asthma. Cochrane Database Syst Rev. 2017 Sep 21;9(9):CD010834. doi: 10.1002/14651858.CD010834.pub3. PMID 28933516
- [Background] MacDonald KM, Kavati A, Ortiz B, Alhossan A, Lee CS, Abraham I. Short- and long-term real-world effectiveness of omalizumab in severe allergic asthma: systematic review of 42 studies published 2008-2018. Expert Rev Clin Immunol. 2019 May;15(5):553-569. doi: 10.1080/1744666X.2019.1574571. Epub 2019 Feb 14. PMID 30763137
- [Background] Papathanassiou E, Loukides S, Bakakos P. Severe asthma: anti-IgE or anti-IL-5? Eur Clin Respir J. 2016 Nov 7;3:31813. doi: 10.3402/ecrj.v3.31813. eCollection 2016. PMID 27834175
- [Background] Ward C, Pais M, Bish R, Reid D, Feltis B, Johns D, Walters EH. Airway inflammation, basement membrane thickening and bronchial hyperresponsiveness in asthma. Thorax. 2002 Apr;57(4):309-16. doi: 10.1136/thorax.57.4.309. PMID 11923548
- [Background] Hsu J, Avila PC, Kern RC, Hayes MG, Schleimer RP, Pinto JM. Genetics of chronic rhinosinusitis: state of the field and directions forward. J Allergy Clin Immunol. 2013 Apr;131(4):977-93, 993.e1-5. doi: 10.1016/j.jaci.2013.01.028. PMID 23540616
- [Background] Chang EH, Willis AL, McCrary HC, Noutsios GT, Le CH, Chiu AG, Mansfield CJ, Reed DR, Brooks SG, Adappa ND, Palmer JN, Cohen NG, Stern DA, Guerra S, Martinez FD. Association between the CDHR3 rs6967330 risk allele and chronic rhinosinusitis. J Allergy Clin Immunol. 2017 Jun;139(6):1990-1992.e2. doi: 10.1016/j.jaci.2016.10.027. Epub 2016 Dec 3. PMID 27923563
- [Background] Kim B, Lee HJ, Im NR, Lee DY, Kim HK, Kang CY, Park IH, Lee SH, Lee HM, Lee SH, Baek SK, Kim TH. Decreased expression of CCL17 in the disrupted nasal polyp epithelium and its regulation by IL-4 and IL-5. PLoS One. 2018 May 10;13(5):e0197355. doi: 10.1371/journal.pone.0197355. eCollection 2018. PMID 29746583
- [Background] Kobayashi N, Terada N, Hamano N, Numata T, Konno A. Transepithelial migration of activated eosinophils induces a decrease of E-cadherin expression in cultured human nasal epithelial cells. Clin Exp Allergy. 2000 Jun;30(6):807-17. doi: 10.1046/j.1365-2222.2000.00827.x. PMID 10848899
- [Background] Steelant B, Seys SF, Van Gerven L, Van Woensel M, Farre R, Wawrzyniak P, Kortekaas Krohn I, Bullens DM, Talavera K, Raap U, Boon L, Akdis CA, Boeckxstaens G, Ceuppens JL, Hellings PW. Histamine and T helper cytokine-driven epithelial barrier dysfunction in allergic rhinitis. J Allergy Clin Immunol. 2018 Mar;141(3):951-963.e8. doi: 10.1016/j.jaci.2017.08.039. Epub 2017 Oct 23. PMID 29074456
- [Background] Hirschberg A, Jokuti A, Darvas Z, Almay K, Repassy G, Falus A. The pathogenesis of nasal polyposis by immunoglobulin E and interleukin-5 is completed by transforming growth factor-beta1. Laryngoscope. 2003 Jan;113(1):120-4. doi: 10.1097/00005537-200301000-00022. PMID 12514394
- [Background] Hakansson K, Bachert C, Konge L, Thomsen SF, Pedersen AE, Poulsen SS, Martin-Bertelsen T, Winther O, Backer V, von Buchwald C. Airway Inflammation in Chronic Rhinosinusitis with Nasal Polyps and Asthma: The United Airways Concept Further Supported. PLoS One. 2015 Jul 1;10(7):e0127228. doi: 10.1371/journal.pone.0127228. eCollection 2015. PMID 26132710
- [Background] Meng J, Zhou P, Liu Y, Liu F, Yi X, Liu S, Holtappels G, Bachert C, Zhang N. The development of nasal polyp disease involves early nasal mucosal inflammation and remodelling. PLoS One. 2013 Dec 10;8(12):e82373. doi: 10.1371/journal.pone.0082373. eCollection 2013. PMID 24340021
- [Background] Tieu DD, Kern RC, Schleimer RP. Alterations in epithelial barrier function and host defense responses in chronic rhinosinusitis. J Allergy Clin Immunol. 2009 Jul;124(1):37-42. doi: 10.1016/j.jaci.2009.04.045. PMID 19560577
- [Background] London NR Jr, Lane AP. Innate immunity and chronic rhinosinusitis: What we have learned from animal models. Laryngoscope Investig Otolaryngol. 2016 Jun;1(3):49-56. doi: 10.1002/lio2.21. Epub 2016 Jun 10. PMID 28459101
- [Background] Van Zele T, Claeys S, Gevaert P, Van Maele G, Holtappels G, Van Cauwenberge P, Bachert C. Differentiation of chronic sinus diseases by measurement of inflammatory mediators. Allergy. 2006 Nov;61(11):1280-9. doi: 10.1111/j.1398-9995.2006.01225.x. PMID 17002703
- [Background] Van Bruaene N, Perez-Novo CA, Basinski TM, Van Zele T, Holtappels G, De Ruyck N, Schmidt-Weber C, Akdis C, Van Cauwenberge P, Bachert C, Gevaert P. T-cell regulation in chronic paranasal sinus disease. J Allergy Clin Immunol. 2008 Jun;121(6):1435-41, 1441.e1-3. doi: 10.1016/j.jaci.2008.02.018. PMID 18423831
- [Background] Terzakis D, Georgalas C. Polyps, asthma, and allergy: what's new. Curr Opin Otolaryngol Head Neck Surg. 2017 Feb;25(1):12-18. doi: 10.1097/MOO.0000000000000323. PMID 27849652
- [Background] Jones AC, Troy NM, White E, Hollams EM, Gout AM, Ling KM, Kicic A, Stick SM, Sly PD, Holt PG, Hall GL, Bosco A. Persistent activation of interlinked type 2 airway epithelial gene networks in sputum-derived cells from aeroallergen-sensitized symptomatic asthmatics. Sci Rep. 2018 Jan 24;8(1):1511. doi: 10.1038/s41598-018-19837-6. PMID 29367592
- [Background] Kanazawa J, Masuko H, Yatagai Y, Sakamoto T, Yamada H, Kaneko Y, Kitazawa H, Iijima H, Naito T, Saito T, Noguchi E, Konno S, Nishimura M, Hirota T, Tamari M, Hizawa N. Genetic association of the functional CDHR3 genotype with early-onset adult asthma in Japanese populations. Allergol Int. 2017 Oct;66(4):563-567. doi: 10.1016/j.alit.2017.02.012. Epub 2017 Mar 17. PMID 28318885
- [Background] Bonnelykke K, Sleiman P, Nielsen K, Kreiner-Moller E, Mercader JM, Belgrave D, den Dekker HT, Husby A, Sevelsted A, Faura-Tellez G, Mortensen LJ, Paternoster L, Flaaten R, Molgaard A, Smart DE, Thomsen PF, Rasmussen MA, Bonas-Guarch S, Holst C, Nohr EA, Yadav R, March ME, Blicher T, Lackie PM, Jaddoe VW, Simpson A, Holloway JW, Duijts L, Custovic A, Davies DE, Torrents D, Gupta R, Hollegaard MV, Hougaard DM, Hakonarson H, Bisgaard H. A genome-wide association study identifies CDHR3 as a susceptibility locus for early childhood asthma with severe exacerbations. Nat Genet. 2014 Jan;46(1):51-5. doi: 10.1038/ng.2830. Epub 2013 Nov 17. PMID 24241537
- [Background] Koppelman GH, Meyers DA, Howard TD, Zheng SL, Hawkins GA, Ampleford EJ, Xu J, Koning H, Bruinenberg M, Nolte IM, van Diemen CC, Boezen HM, Timens W, Whittaker PA, Stine OC, Barton SJ, Holloway JW, Holgate ST, Graves PE, Martinez FD, van Oosterhout AJ, Bleecker ER, Postma DS. Identification of PCDH1 as a novel susceptibility gene for bronchial hyperresponsiveness. Am J Respir Crit Care Med. 2009 Nov 15;180(10):929-35. doi: 10.1164/rccm.200810-1621OC. Epub 2009 Sep 3. PMID 19729670
- [Background] Kozu Y, Gon Y, Maruoka S, Kazumichi K, Sekiyama A, Kishi H, Nomura Y, Ikeda M, Hashimoto S. Protocadherin-1 is a glucocorticoid-responsive critical regulator of airway epithelial barrier function. BMC Pulm Med. 2015 Jul 31;15:80. doi: 10.1186/s12890-015-0078-z. PMID 26227965
- [Background] Post S, Heijink IH, Hesse L, Koo HK, Shaheen F, Fouadi M, Kuchibhotla VNS, Lambrecht BN, Van Oosterhout AJM, Hackett TL, Nawijn MC. Characterization of a lung epithelium specific E-cadherin knock-out model: Implications for obstructive lung pathology. Sci Rep. 2018 Sep 5;8(1):13275. doi: 10.1038/s41598-018-31500-8. PMID 30185803
- [Background] Masuyama K, Morishima Y, Ishii Y, Nomura A, Sakamoto T, Kimura T, Mochizuki M, Uchida Y, Sekizawa K. Sputum E-cadherin and asthma severity. J Allergy Clin Immunol. 2003 Jul;112(1):208-9. doi: 10.1067/mai.2003.1526. No abstract available. PMID 12847501
- [Background] Ierodiakonou D, Postma DS, Koppelman GH, Boezen HM, Gerritsen J, Ten Hacken N, Timens W, Vonk JM. E-cadherin gene polymorphisms in asthma patients using inhaled corticosteroids. Eur Respir J. 2011 Nov;38(5):1044-52. doi: 10.1183/09031936.00194710. Epub 2011 May 3. PMID 21540309
- [Background] Wang MF, Kuo SH, Huang CH, Chen YJ, Lin SH, Lee CJ, Lue KH, Wu SC, Cho CY, Wong RH. Exposure to environmental tobacco smoke, human E-cadherin C-160A polymorphism, and childhood asthma. Ann Allergy Asthma Immunol. 2013 Oct;111(4):262-7. doi: 10.1016/j.anai.2013.07.008. Epub 2013 Aug 2. PMID 24054361
- [Background] Fitzpatrick AM, Moore WC. Severe Asthma Phenotypes - How Should They Guide Evaluation and Treatment? J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):901-908. doi: 10.1016/j.jaip.2017.05.015. PMID 28689840
- [Background] Rasmussen F, Taylor DR, Flannery EM, Cowan JO, Greene JM, Herbison GP, Sears MR. Risk factors for airway remodeling in asthma manifested by a low postbronchodilator FEV1/vital capacity ratio: a longitudinal population study from childhood to adulthood. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1480-8. doi: 10.1164/rccm.2108009. PMID 12045120
- [Background] Chae EJ, Kim TB, Cho YS, Park CS, Seo JB, Kim N, Moon HB. Airway Measurement for Airway Remodeling Defined by Post-Bronchodilator FEV1/FVC in Asthma: Investigation Using Inspiration-Expiration Computed Tomography. Allergy Asthma Immunol Res. 2011 Apr;3(2):111-7. doi: 10.4168/aair.2011.3.2.111. Epub 2010 Dec 1. PMID 21461250
- [Background] Inoue H, Ito I, Niimi A, Matsumoto H, Matsuoka H, Jinnai M, Takeda T, Oguma T, Otsuka K, Nakaji H, Tajiri T, Iwata T, Nagasaki T, Kanemitsu Y, Mishima M. CT-assessed large airway involvement and lung function decline in eosinophilic asthma: The association between induced sputum eosinophil differential counts and airway remodeling. J Asthma. 2016 Nov;53(9):914-21. doi: 10.3109/02770903.2016.1167903. Epub 2016 Apr 26. PMID 27115448
- [Background] Saglani S, Lloyd CM. Novel concepts in airway inflammation and remodelling in asthma. Eur Respir J. 2015 Dec;46(6):1796-804. doi: 10.1183/13993003.01196-2014. Epub 2015 Nov 5. PMID 26541520
- [Background] Castro-Rodriguez JA, Saglani S, Rodriguez-Martinez CE, Oyarzun MA, Fleming L, Bush A. The relationship between inflammation and remodeling in childhood asthma: A systematic review. Pediatr Pulmonol. 2018 Jun;53(6):824-835. doi: 10.1002/ppul.23968. Epub 2018 Feb 22. PMID 29469196
- [Background] Davies DE. Epithelial barrier function and immunity in asthma. Ann Am Thorac Soc. 2014 Dec;11 Suppl 5:S244-51. doi: 10.1513/AnnalsATS.201407-304AW. PMID 25525727
- [Background] Holgate ST. Epithelium dysfunction in asthma. J Allergy Clin Immunol. 2007 Dec;120(6):1233-44; quiz 1245-6. doi: 10.1016/j.jaci.2007.10.025. PMID 18073119
- [Background] Laitinen LA, Heino M, Laitinen A, Kava T, Haahtela T. Damage of the airway epithelium and bronchial reactivity in patients with asthma. Am Rev Respir Dis. 1985 Apr;131(4):599-606. doi: 10.1164/arrd.1985.131.4.599. PMID 3994155
- [Background] Qin L, Gibson PG, Simpson JL, Baines KJ, McDonald VM, Wood LG, Powell H, Fricker M. Dysregulation of sputum columnar epithelial cells and products in distinct asthma phenotypes. Clin Exp Allergy. 2019 Nov;49(11):1418-1428. doi: 10.1111/cea.13452. Epub 2019 Aug 6. PMID 31264263